CLINICAL TRIAL: NCT06517095
Title: Revised Capsular Polishing and Its Impact on the Positioning of the Intraocular Lens and Visual Quality Following Femtosecond Laser-assisted Cataract Surgery
Acronym: ELPVQFLACS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Conflict of interest
Sponsor: Xi'an People's Hospital (Xi'an Fourth Hospital) (Other)
Responsible Party: Principal Investigator, Xin Zhou, Associate Senior Doctor, Xi'an People's Hospital (Xi'an Fourth Hospital)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20150824
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Cataract
Keywords: visual acuity; visual quality; polishing; femtosecond laser
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: The intervening measure is utilize the OVDs to partially fill the peripheral capsule, causing the central posterior capsule to bulge, and then employ the double-ended Whitman Shepherd capsular polisher to meticulously polish both the anterior and equator of the capsule. By rotating the polisher 180°along one side, followed by switching ends to cover the remaining 180° range, even the main incision site can be effectively addressed due to its curved tip design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polished (Active Comparator): The polished group did the improved capsular polishing.
  Interventions: Procedure: improved capsular polishing
- control (Placebo Comparator): The control group did not undergo improved polishing, the conventional I/A polishing the capsule instead.
  Interventions: Procedure: the conventional I/A polishing

INTERVENTIONS:
Procedure: improved capsular polishing — In the polished group,utilize the OVDs to partially fill the peripheral capsule, causing the central posterior capsule to bulge, and then employ the double-ended Whitman Shepherd capsular polisher to meticulously polish both the anterior and equator of the capsule. This process also allows for simultaneous polishing of a portion of the posterior capsule. By rotating the polisher 180°along one side, followed by switching ends to cover the remaining 180° range, even the main incision site can be effectively addressed due to its curved tip design.
  Arms: polished
Procedure: the conventional I/A polishing — the conventional I/A polishing the capsule
  Arms: control

SUMMARY:
This study aims to investigate the impact of improved capsular polishing on the long-term stability of effective lens position (ELP) and visual quality in patients following femtosecond laser-assisted cataract surgery combined with intraocular lens implantation. Throughout the follow-up period, changes in ELP were observed using OCT to measure the central corneal posterior surface to the IOL anterior surface. The contraction of the anterior capsule orifice was assessed through anterior segment photography, and its diameter and area were measured and analyzed using drawing software at each follow-up visit. Additionally, the investigators analyzed the correlation between the degree of anterior capsule orifice contraction and ELP, as well as examined whether ACO formed and its degree, PCO formation and its degree. Objective examination using OQAS II was conducted to measure PSF, MTF, OSI, and SR of patients; high-order aberrations including astigmatism, trifolium, and spherical aberration were measured by OPD-Scan III. Furthermore, the investigators investigated the correlation between ACO/PCO degrees and visual quality.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with age-related cataract
2. Patients seeking to reduce their reliance on corrective eyewear postoperative and exhibiting high expectations for optimal visual acuity at all distances - near, intermediate, and distant
3. Anticipated postoperative astigmatism of ≤1.00D
4. Pupil diameter in a darkened environment ranging from 3.0-5.5 mm
5. Kappa angle ≤0.5 mm or less than half the diameter of the central refractive optical zone of the MIOL.

Exclusion Criteria:

1. Progressive and aggravated retinal diseases, such as diabetic retinopathy, macular degeneration, preretinal membrane, vitreous macular traction syndrome, Stargardt disease, retinitis pigmentosa, etc., and serious optic nerve diseases
2. Small eyeballs, ultra-high myopia, obvious pupil abnormalities, severe corneal lesions, severe irregular astigmatism, chronic uveitis, glaucoma, obvious abnormalities of lens capsule membrane and suspension ligament, major degree alternating strabismus and other ocular organic diseases and amblyopia
3. Severe mental and psychological diseases
4. History of internal eye surgery
5. Posterior capsule rupture or uneventful in-the-bag IOL implantation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
visual acuity | The data were collected at various time points for follow-up: preoperative, 1-day postoperative, 1-week postoperative, 1-month postoperative, 3-month postoperative, 6-month postoperative, and 1-year postoperative.
  Utilize decimal visual acuity charts for assessment purposes and record the findings in LogMAR format to facilitate statistical analysis.
strehl ratio(SR) | The data were collected at various time points for follow-up: preoperative, 1-day postoperative, 1-week postoperative, 1-month postoperative, 3-month postoperative, 6-month postoperative, and 1-year postoperative.
  This is one of the visual quality indicators. It's assessed by OQAS II instrument. SR that represents the ratio of the central peak value of the point spread function in an aberration-free system to that in a aberration system with the same pupil diameter, the higher the value is, the better the optical quality is.
modulation transfer function cutoff frequency (MTF cutoff) | The data were collected at various time points for follow-up: preoperative, 1-day postoperative, 1-week postoperative, 1-month postoperative, 3-month postoperative, 6-month postoperative, and 1-year postoperative.
  MTF cutoff that characterizes the spatial frequency corresponding to the minimum resolution of human eyes in the modulation transfer function curve, and the higher the value is, the better the optical quality becomes,and it is immune to subjective factors and provides an objective assessment of the optical imaging quality across the entire refractive system of the artificial lens eye.
objective scatter index (OSI) | The data were collected at various time points for follow-up: preoperative, 1-day postoperative, 1-week postoperative, 1-month postoperative, 3-month postoperative, 6-month postoperative, and 1-year postoperative.
  OSI that objectively reflects the scatter of the refractive medium,a higher OSI ratio indicates a more severe degree of scatter in the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Xin Zhou, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No